CLINICAL TRIAL: NCT06506110
Title: Determining the Patient Acceptable Symptom State (PASS) for Acute Pain After Surgery - A Retrospective Study
Brief Title: PASS Pain After Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5290; CAPCR# 24-5290 (Other: UHN)
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Analgesia
Keywords: PASS; MCID; NRS pain score; Acute pain
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received intravenous PCA following surgery at the UHN: Patients who received intravenous PCA following surgery at the UHN from the period of June 4, 2022 to December 31, 2023.
  Interventions: Other: Retrieving of retrospective data from Epic

INTERVENTIONS:
Other: Retrieving of retrospective data from Epic — Retrospective data from Epic will be extracted to determine the Patient Acceptable Symptom State (PASS) for the numeric rating scale (NRS) pain score in the first 48 hours after surgery in patients who received intravenous Patient Controlled Analgesia.

SUMMARY:
The numeric rating scale (NRS) is one way to assess how much pain a patient is feeling after surgery, ranging from 0 (no pain) to 10 (the worst pain imaginable). The score getting lower can thus indicate pain relief. However, a small change in the score does not mean that the patient is actually satisfied with their pain relief treatment. The PASS (patient acceptable symptom state) is the score threshold beyond which a patient considers their treatment satisfactory.

The purpose of this observational study is to find out the PASS for the NRS in the first 48 hours after surgery. This will help guide future research on pain medicine, so that new techniques can deliver adequate patient satisfaction.

DETAILED DESCRIPTION:
As healthcare delivery and research studies become more patient-centered, patient-reported outcome measures (PROMs) - instruments completed by a patient to capture their health status (e.g., pain, quality of life, function) - are increasingly used. However little attention has been paid to PROMs in the acute phase of postoperative recovery. Given that many patients experience moderate to severe pain in the first day following surgery (e.g., 50% for joint replacement surgery), and that acute postsurgical pain is associated with long-term outcomes, a focus on patient-reported acute pain following surgery is needed.

Both acute and chronic postoperative pain are commonly assessed using the 100 mm visual analogue scale (VAS, 0 mm = no pain to 100 mm = worst possible pain) or numeric rating scale (NRS, 0 = no pain to 10 = worst possible pain). While a reduction in the VAS or NRS pain score indicates some degree of pain relief, neither the raw numerical score nor the statistical significance of a score's change indicates whether the change is perceived by patients to be meaningful. Instead, the Patient Acceptable Symptom State (PASS), which represents the threshold beyond which patients consider themselves well or satisfied with a treatment, can be used to determine the proportion of patients that responded to treatment (i.e., the proportion of patients that achieved the PASS) and to calculate the number needed to treat. Little to no data has been found concerning the PASS for acute postsurgical pain. There has been somewhat more work quantifying the Minimum Clinically Important Difference (MCID; the smallest change that is important to patients), which is a related concept to the PASS that also determines the clinical significance of a change in pain score. The MCID varies widely across chronic pain disorders (from 8 mm for scleroderma to 82 mm for trigeminal neuralgia) and across non-surgical acute pain conditions (from 8 mm for patients presenting to the emergency department to 40 mm for rheumatic conditions). Therefore, the PASS for acute pain following surgeries is expected to vary based on the type of surgery, but this has not been determined. Similarly, there is no known study of the consistency in PASS throughout the postoperative period or across the patient and surgical factors that are known to be important for MCID (e.g., preoperative pain, pain expectations), or the opioid dose (measured in morphine milligram equivalents) needed to achieve the PASS.

The primary objective of this study is to determine the PASS for the NRS pain score in the first 48 hours after surgery in patients who received intravenous patient-controlled analgesia (PCA). The study includes patients who have undergone surgery at UHN between June 4, 2022, and December 31, 2023 (the study period). Patients will be identified using the Epic data management software. All required data for this study will be obtained from the Epic electronic medical record at UHN. For patients who are on intravenous PCA, the patient's pain score at rest and with activity is taken using the NRS multiple times per day and recorded in Epic. Each time the NRS is taken, the patient's satisfaction (yes/no) is also recorded along with the cumulative PCA opioid dose.

This study will include a descriptive analysis of the data collected. The descriptive analysis will be used to summarize the characteristics of the study population and to identify patterns and trends in the data. Measures of central tendency (e.g., mean, median, mode) and measures of variability (e.g., standard deviation, range) will be calculated for continuous variables. Frequency distributions and proportions will be used to describe categorical variables. Missing data will not be imputed but will be reported for every variable. Graphs and charts will be used to visualize the data. Histograms, bar charts, and pie charts will be used to describe the distribution of continuous and categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Had surgery at the UHN during the study period
* Received intravenous PCA within the first 48 hours after surgery
* Have at least 1 NRS rating and 1 satisfaction rating in the first 48 hours after surgery

Exclusion Criteria:

* Use of epidural analgesia in the first 48 hours after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who received intravenous patient-controlled analgesia (PCA) following surgery at the University Health Network (UHN) during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
PASS for the NRS | First 48 hours after surgery
  The PASS for the NRS pain score in the first 48 hours after surgery in patients who received intravenous PCA.
  To determine PASS, patients responding "yes" to the satisfaction question in Epic are considered to have an acceptable pain state at that time. Each patient can contribute multiple NRS scores. PASS will be calculated as:
  * the 75th centile of the NRS taken at the time of the "yes" satisfaction response
  * the highest NRS pain score at which each patient considers themselves satisfied. The NRS PASS will be the mean of these scores.
  * the NRS cut-off that optimizes the sensitivity and specificity between satisfied and unsatisfied responses using receiver-operating characteristic (ROC) curves
  The method that gives the PASS with the best sensitivity and specificity will be determined. These methods will be used to calculate the PASS separately for pain at rest and with movement. This will be done for the entire 48-hour period, separately for each surgery.

SECONDARY OUTCOMES:
Consistency of PASS for the NRS | First 48 hours after surgery
  The degree to which the PASS for the NRS pain score changes across the PACU, and the first 0-6, 6-12, 12-24, 24-36, and 36-48 hours after surgery, separately for each surgery.
Patient and procedure factors associated with PASS for the NRS | First 48 hours after surgery
  To determine the patient and procedure factors associated with the PASS, a subgroup analysis will be conducted to explore differences in the PASS (with a 95% confidence interval) for different patient groups (e.g., preoperative use of opioids, sex, age, comorbidities). Descriptive statistics and graphical representations will be used for each subgroup. Factors associated with the PASS will be explored using multivariable models (which may include logistic regression, Poisson regression, negative binomial regression, according to the nature of the data) adjusting for patient and procedure characteristics. Tests will be 2-sided and a p-value less than 0.05 will be considered statistically significant.
Opioid dose needed to achieve PASS for the NRS | First 48 hours after surgery
  To determine the opioid dose (in morphine milligram equivalents) that is required to achieve the PASS for the NRS, the median opioid dose in the 4 hours before the NRS was taken will be calculated for those patients that achieved the PASS (with 95% confidence interval). It will be explored whether this varies by patient and procedure factors.
MCID for the NRS | First 48 hours after surgery
  The MCID for the NRS pain score in the first 48 hours after surgery in patients who received intravenous PCA.
  Distribution-based methods will be used to determine the MCID for the NRS. The MCID will be defined as:
  * 0.3 standard deviations of the NRS pain scores taken in the first 48 hours after surgery
  * The Standard Error of the Measurement (SEM) of NRS pain scores taken in the first 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laura Giron-Arango, MD, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No